CLINICAL TRIAL: NCT03121352
Title: Pilot Study of Carboplatin, Nab-Paclitaxel and Pembrolizumab for Metastatic Triple-Negative Breast Cancer
Brief Title: Carboplatin, Nab-Paclitaxel and Pembrolizumab for Metastatic Triple-Negative Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Joseph Baar, MD, PhD, Associate Professor of Medicine, Case Comprehensive Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE6115
Record Dates: First submitted 2017-03-30; First posted 2017-04-20 (Actual); Results first posted 2023-10-06 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-10

CONDITIONS: Metastatic Triple Negative Breast Cancer
Keywords: Carboplatin; Nab-Paclitaxel; Pembrolizumab
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — Carboplatin; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Carboplatin + Nab-paclitaxel + Pembrolizumab (Experimental): Combination therapy of Carboplatin, Nab-paclitaxel, and Pembrolizumab
  Interventions: Drug: Carboplatin; Drug: Nab-paclitaxel; Drug: Pembrolizumab

INTERVENTIONS:
Drug: Carboplatin — AUC 4.5 IV day 1 of 21-day cycle
Drug: Nab-paclitaxel — 75mg/m2 IV days 1, 8 and 15 of 21-day cycle
  Other Names: Abraxane
Drug: Pembrolizumab — 200 mg IV every 21 days
  Other Names: MK-3475

SUMMARY:
The purpose of this study is to see how effective the combination of the two chemotherapy drugs (carboplatin and nab-paclitaxel) are when added to a third drug, pembrolizumab.

Pembrolizumab is an investigational (experimental) drug that works by reinvigorating the immune system, allowing it to target and destroy cancer cells. Pembrolizumab is experimental because it is not approved by the Food and Drug Administration (FDA) for this type of breast cancer treatment.

DETAILED DESCRIPTION:
Primary Objective - Determine overall response rate (ORR) in patients treated with CNP

Secondary Objective(s)

* Determine progression-free survival (PFS), and disease control rate (DCR) in patients treated with CNP.
* Determine duration of response in patients treated with CNP.
* Determine safety/tolerability of CNP.

Correlative Endpoints

- Identify pathologic and genomic correlates of response to CNP.

Study design including dose escalation / cohorts This is prospective pilot clinical trial of CNP in up to 30 patients with mTNBC

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have histologically or cytologically confirmed metastatic triple negative breast cancer
* Subjects must have received no more than 2 prior therapies for this disease
* ECOG Performance Status 0-1
* Subjects must have normal organ and marrow function as defined below:

  * Hemoglobin ≥ 10.0 g/dl
  * Absolute neutrophil count ≥ 1,000/μL
  * Platelet count ≥ 100,000/μL
  * Total bilirubin within normal institutional limits
  * AST (SGOT) ≤ 2.5 X institutional upper limit of normal
  * ALT (SGPT) ≤ 2.5 X institutional upper limit of normal
  * Serum creatinine ≤ 1.5 normal institutional limits
* Life expectancy of 12 weeks or more
* Subjects must have the ability to understand and the willingness to sign a written informed consent document
* Subjects must have measurable disease per RECIST v1.1
* Subjects must be willing to undergo a preliminary biopsy of a metastatic focus for research purposes. A second post-treatment biopsy will be offered but will not be mandated

Exclusion Criteria:

* Prior treatment toxicities have not resolved to ≤ Grade 1 according to NCI CTCAE Version 4.0 (except for alopecia and neuropathy)
* Subjects receiving any other investigational agents
* Subjects with radiographically stable treated brain metastases are eligible but must not have been on steroid therapy for at least 4 weeks
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to nab-paclitaxel, carboplatin, pembrolizumab, or other agents used in this study
* Subjects with uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant or breastfeeding women are excluded from this study
* Patients with conditions requiring immunosuppressive medications or chronic infections (including HIV infection, hepatitis B and C)
* Patients with chronic autoimmune disease
* Patients with prior therapy with antibodies that modulate T-cell function (e.g., anti-PD-1, anti-PD-L1)
* Patients with evidence of active, non-infectious pneumonia
* Patients active infection requiring intravenous systemic therapy
* Patients with known psychiatric or substance abuse disorders that would interfere with cooperation with requirements of the trial
* Patients who have received a live vaccine within 30 days prior to the first dose of pembrolizumab
* Patients with a known additional malignancy that is progressing or requires active treatment (within the last 5 years). Exceptions: basal cell carcinoma of the skin, squamous cell carcinoma of the skin or in situ cervical cancer that has undergone potentially curative therapy
* Patients who have received monoclonal anti-cancer antibody within 4 weeks of first dose of study drugs
* Patients who have received chemotherapy, small molecule targeted therapy or radiation within the 2 weeks of first dose of study drugs
* Patients who have participated in MK-3475 Merck studies
* Patients with carcinomatous meningitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-05-19 (Actual); Primary Completion 2022-02-20 (Actual); Study Completion 2022-05-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Baar, MD, Principal Investigator — University Hospitals Cleveland Medical Center, Seidman Cancer Center, Case Comprehensive Cancer Center
Locations (2):
- United States (2):
  - University Hospitals Cleveland Medical Center, Seidman Cancer Center, Case Comprehensive Cancer Center, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center, Cleveland, Ohio

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Carboplatin + Nab-paclitaxel + Pembrolizumab
Started | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Carboplatin + Nab-paclitaxel + Pembrolizumab
Number analyzed (Participants) | 30
Age, Customized [Number; unit: participants]
  30-39 years | 2
  40-49 years | 7
  50-59 years | 11
  60-69 years | 4
  70-79 years | 5
  80-89 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 30
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 24
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR) in Patients Treated With CNP
Description: The number of people with tumor responses according to RECIST (V1.1). These responses include Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. Progressive Disease (PD): At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progression). Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study
Time Frame: Up to 24 months
Population: All participants who were evaluable for clinical response. Three participants were not evaluable for treatment response per Principal Investigator's assessment
Measure: Count of Participants; unit: Participants
Arm/Group | Carboplatin + Nab-paclitaxel + Pembrolizumab
Number analyzed (Participants) | 27
Participants
  Complete Response (CR) | 2
  Partial Response (PR) | 11
  Progressive Disease (PD) | 6
  Stable Disease (SD) | 8

2. Secondary Outcome: Progression-free Survival (PFS) in Patients Treated With CNP
Description: Average time (in months) patient's tumors did not progress according to the RECIST criteria (V1.1). Progressive disease is defined as Progressive Disease (PD): At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm
Time Frame: Up to 24 months
Population: All participants who received treatment.
Measure: Mean (95% Confidence Interval); unit: months
Arm/Group | Carboplatin + Nab-paclitaxel + Pembrolizumab
Number analyzed (Participants) | 30
months | 5.8 [4.7 to 8.5]

3. Secondary Outcome: Disease Control Rate (DCR) in Patients Treated With CNP
Description: the percentage of patients with advanced or metastatic cancer who have achieved complete response, partial response and stable disease to a therapeutic intervention. Responses are defined as Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm or Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study
Time Frame: Up to 24 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Carboplatin + Nab-paclitaxel + Pembrolizumab
Number analyzed (Participants) | 27
Participants | 21

4. Secondary Outcome: Duration of Response in Patients Treated With CNP
Description: Average time patients have a response, as defined by the RECIST criteria (V1.1). Response includes: Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm or Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: Up to 24 months
Population: Participants who have a CR and PR response from treatment
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Carboplatin + Nab-paclitaxel + Pembrolizumab
Number analyzed (Participants) | 13
Months
  Complete: number analyzed (Participants) | 2
  Complete | NA [NA to NA] — The median duration for complete response was not reached. The two patients who had a complete response never progressed during the entire time of the study, and therefore, their response was ongoing at the time of the data analysis.
  Partial: number analyzed (Participants) | 11
  Partial | 6.3 [3 to 7]

ADVERSE EVENTS:
Time Frame: Up to five years after cycle six of treatment
Arm/Group | Carboplatin + Nab-paclitaxel + Pembrolizumab
All-Cause Mortality (participants affected / at risk) | 27/30
Serious Adverse Events (participants affected / at risk) | 13/30
Other Adverse Events (participants affected / at risk) | 30/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Carboplatin + Nab-paclitaxel + Pembrolizumab (N=30)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Severe Left Thigh Pain Due to a Hematoma (Musculoskeletal and connective tissue disorders) | 1 (1)
Creatinine increased (Investigations) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Breast infection (Infections and infestations) | 1 (2)
Fever (General disorders) | 2 (2)
INR increased (Blood and lymphatic system disorders) | 1 (1)
Alanine aminotransferase increased (Investigations) | 2 (2)
Autoimmune disorder-hepatitis (Immune system disorders) | 1 (1)
Lung infection (pneumonia) (Infections and infestations) | 2 (2)
Urinary tract infection (Infections and infestations) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Device related infection (Infections and infestations) | 1 (2)
Soft tissue infection (Infections and infestations) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Death due to disease progression (General disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1)
Psychosis-altered mental status (Psychiatric disorders) | 1 (1)
Infection (Infections and infestations) | 1 (3)
Allergic reaction (Immune system disorders) | 1 (1)
Generalized pain-hip and lower extremities (Musculoskeletal and connective tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Carboplatin + Nab-paclitaxel + Pembrolizumab (N=30)
Abdominal pain (Gastrointestinal disorders) | 3 (6)
Acute kidney injury (Renal and urinary disorders) | 1 (3)
Alanine aminotransferase increased (Investigations) | 8 (19)
Alkaline phosphatase increased (Investigations) | 4 (4)
Allergic reaction (Immune system disorders) | 2 (3)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Alopecia (Skin and subcutaneous tissue disorders) | 20 (39)
Anal pain (Gastrointestinal disorders) | 1 (2)
Anemia (Blood and lymphatic system disorders) | 21 (109)
Anorexia (Metabolism and nutrition disorders) | 15 (25)
Anxiety (Psychiatric disorders) | 6 (13)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (3)
Aspartate aminotransferase increased (Investigations) | 6 (19)
Ataxia (Nervous system disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (5)
Bloating (Gastrointestinal disorders) | 1 (1)
Iron Deficiency (Blood and lymphatic system disorders) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1)
Blurred vision (Eye disorders) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Breast infection (Infections and infestations) | 1 (1)
Breast pain (Reproductive system and breast disorders) | 5 (6)
Bronchial infection (Infections and infestations) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 1 (1)
Buttock pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Carbon monoxide diffusing capacity decreased (Investigations) | 1 (1)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Confusion (Psychiatric disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 13 (19)
Cough (Respiratory, thoracic and mediastinal disorders) | 9 (15)
Creatinine increased (Investigations) | 4 (15)
Death NOS (General disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 3 (5)
Depression (Psychiatric disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 18 (38)
Dizziness (Nervous system disorders) | 7 (11)
Dry eye (Eye disorders) | 2 (2)
Dry mouth (Gastrointestinal disorders) | 3 (3)
Dry skin (Skin and subcutaneous tissue disorders) | 3 (3)
Dysgeusia (Nervous system disorders) | 10 (13)
Dyspepsia (Gastrointestinal disorders) | 2 (6)
Dysphasia (Nervous system disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 9 (18)
Edema limbs (General disorders) | 6 (7)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Erythroderma (Skin and subcutaneous tissue disorders) | 1 (6)
Blood shot eyes, capillary ruptures intermittently (Eye disorders) | 1 (1)
Aura, intermittent (Eye disorders) | 1 (1)
Scleral disease (Eye disorders) | 1 (1)
Visitoin - aura (intermittent) (Eye disorders) | 1 (1)
Red sclera (Eye disorders) | 1 (1)
Facial muscle weakness (Nervous system disorders) | 1 (1)
Facial pain (General disorders) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 3 (7)
Fatigue (General disorders) | 17 (56)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Flu like symptoms (General disorders) | 1 (1)
Flushing (Vascular disorders) | 2 (4)
Fracture (Injury, poisoning and procedural complications) | 1 (1)
Broken tooth (Gastrointestinal disorders) | 1 (1)
Heartburn (Gastrointestinal disorders) | 1 (1)
Elevated Vitamin D (General disorders) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 7 (17)
Gingival pain (Gastrointestinal disorders) | 1 (1)
Headache (Nervous system disorders) | 6 (8)
Hot flashes (Vascular disorders) | 5 (5)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (2)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 3 (3)
Hyperkalemia (Metabolism and nutrition disorders) | 3 (5)
Hypernatremia (Metabolism and nutrition disorders) | 3 (4)
Hypertension (Vascular disorders) | 6 (12)
Hyperthyroidism (Endocrine disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 7 (7)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (10)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 9 (23)
Hypomagnesemia (Metabolism and nutrition disorders) | 13 (30)
Hyponatremia (Metabolism and nutrition disorders) | 7 (12)
Hypotension (Vascular disorders) | 4 (6)
Hypothyroidism (Endocrine disorders) | 7 (7)
Immune related hepatitis (Immune system disorders) | 1 (1)
Infection-other (Infections and infestations) | 1 (1)
Infusion related reaction (General disorders) | 2 (2)
Insomnia (Psychiatric disorders) | 4 (9)
Lymphedema (Vascular disorders) | 1 (1)
Lymphocyte count decreased (Investigations) | 11 (65)
Mucositis oral (Gastrointestinal disorders) | 4 (4)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3)
Nail discoloration (Skin and subcutaneous tissue disorders) | 3 (3)
Nail infection (Infections and infestations) | 1 (1)
Nail loss (Skin and subcutaneous tissue disorders) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 20 (42)
Neck edema (General disorders) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Aura, intermittent (Nervous system disorders) | 1 (1)
Heat sensation, lower right back (Nervous system disorders) | 1 (1)
Neutrophil count decreased (Investigations) | 20 (91)
Non-cardiac chest pain (General disorders) | 4 (4)
Oral pain (Gastrointestinal disorders) | 1 (1)
Otitis media (Infections and infestations) | 1 (1)
Pain (General disorders) | 9 (10)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (4)
Pain of skin (Skin and subcutaneous tissue disorders) | 2 (2)
Papulopustular rash (Infections and infestations) | 2 (2)
Pelvic pain (Reproductive system and breast disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 12 (27)
Platelet count decreased (Investigations) | 15 (54)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Presyncope (Nervous system disorders) | 2 (2)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (5)
Psychosis (Psychiatric disorders) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (2)
Rash pustular (Infections and infestations) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 6 (6)
Sinusitis (Infections and infestations) | 3 (5)
Blistering, left leg (Skin and subcutaneous tissue disorders) | 1 (1)
Facial redness/bumpy/moon face (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Spasticity (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Tooth infection (Infections and infestations) | 1 (1)
Tremor (Nervous system disorders) | 1 (1)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Upper respiratory infection (Infections and infestations) | 2 (2)
Urinary frequency (Renal and urinary disorders) | 1 (1)
Urinary tract infection (Infections and infestations) | 4 (5)
Vertigo (Ear and labyrinth disorders) | 1 (2)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 9 (12)
Watering eyes (Eye disorders) | 1 (1)
Weight gain (Investigations) | 1 (1)
Weight loss (Investigations) | 7 (10)
White blood cell decreased (Investigations) | 21 (137)
Wound infection (Infections and infestations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-04-04): https://cdn.clinicaltrials.gov/large-docs/52/NCT03121352/Prot_SAP_000.pdf
  • Informed Consent Form (2022-03-23): https://cdn.clinicaltrials.gov/large-docs/52/NCT03121352/ICF_001.pdf